CLINICAL TRIAL: NCT06146049
Title: Examination of Participation Trends and Engagement Patterns of Participants in Post Traumatic Stress Disorder Clinical Trials
Brief Title: Exploring Clinical Study Experiences of People With Post Traumatic Stress Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 65314844
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in post traumatic stress disorder observational study serves as a crucial contribution to advancing medical knowledge and refining the care provided to individuals facing similar health challenges.

The primary objective centers on a meticulous examination of trial completion rates and voluntary withdrawals within this distinct patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of post traumatic stress disorder
* No prior treatment for post traumatic stress disorder
* Willing and able to provide informed consent.

Exclusion Criteria:

* Enrolled in another research study
* Psychiatric or behavioral illness
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post traumatic stress disorder patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a post traumatic stress disorder clinical research. | 3 months
Number of post traumatic stress disorder study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casarin J, Ielmini M, Cromi A, Lagana AS, Poloni N, Callegari C, Ghezzi F. Post-traumatic stress following total hysterectomy for benign disease: an observational prospective study. J Psychosom Obstet Gynaecol. 2022 Mar;43(1):11-17. doi: 10.1080/0167482X.2020.1752174. Epub 2020 Apr 22. PMID 32319346
- [Background] Lai X, Chen J, Li H, Zhou L, Huang Q, Liao Y, Krewski D, Wen SW, Zhang L, Xie RH. The incidence of post-traumatic stress disorder following traumatic childbirth: A systematic review and meta-analysis. Int J Gynaecol Obstet. 2023 Jul;162(1):211-221. doi: 10.1002/ijgo.14643. Epub 2023 Jan 19. PMID 36571476
- [Background] Cenkner DP, Asnaani A, DiChiara C, Harb GC, Lynch KG, Greene J, Scott JC. Neurocognitive Predictors of Treatment Outcomes in Cognitive Processing Therapy for Post-traumatic Stress Disorder: Study Protocol. Front Psychol. 2021 Jan 26;12:625669. doi: 10.3389/fpsyg.2021.625669. eCollection 2021. PMID 33574791

DOCUMENTS (1):
  • Informed Consent Form (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT06146049/ICF_000.pdf